CLINICAL TRIAL: NCT05328726
Title: A Double-blind, Randomized, Placebo-controlled, Sequential, Single, Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Parameters of Subcutaneous Injections of GZR18 in Healthy Subjects
Brief Title: Single, Ascending Dose, First Time in Human Study for GZR18 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-1012
Record Dates: First submitted 2022-02-25; First posted 2022-04-14 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, randomized, placebo-controlled, sequential, dose-escalating, single-dose study.
Who Masked: Participant, Investigator
Masking Description: Enrollment of up to 56 subjects in up to 7 cohorts may occur. Randomization is 3:1 (active drug:placebo) across all cohorts. Within each cohort, 6 subjects will be randomized to receive GZR18, and 2 subjects will be randomized to receive placebo.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug:GZR-18 administered via subcutaneous injection (Experimental): For Assigned Interventions: GZR-18 administered once via subcutaneous injection at doses of 1.0 ug/kg, 5.0 ug/kg, 10.0 ug/kg, 20.0 ug/kg, 30.0 ug/kg, 40.0 ug/kg & 50.0 ug/kg
  Interventions: Drug: GZR-18
- Placebo control (Placebo Comparator): Commercially obtained sterile, normal saline for injection will be used as the matching placebo. Placebo will be dosed in an identical manner to active study drug. The volume of placebo will be calculated according to body weight using active drug dose for volume calculation in order to maintain the study blind.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR-18 — As previously described in Arms
  Arms: Drug:GZR-18 administered via subcutaneous injection
Other: Placebo — Placebo will be dosed in an identical manner to active study drug.
  Other Names: Placebo Control
  Arms: Placebo control

SUMMARY:
Single ascending dose first time in human study for GZR18 in healthy subjects

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, sequential, single, ascending dose study to evaluate the safety, tolerability, pharmacokinetic, and pharmacodynamic parameters of subcutaneous injections of GZR18 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date informed consent prior to any study-related activities being performed
2. Be considered healthy in the opinion of the PI or qualified designee and have no clinically significant abnormal laboratory values at screening
3. Male
4. Aged 18 to 60 years, inclusive, at the time of signing the informed consent. Note: if the study is to be conducted at a clinical site located in Lincoln, Nebraska, the lower age limit will be 19 years of age
5. Have a BMI between 20.0 to 35.0 kg/m2, inclusive, at Screening or check-in prior to dosing
6. Have a normal renal function as defined by estimated glomerular filtration rate (eGFR) > 90 mL/min/1.73m2 at Screening or check-in prior to dosing
7. Be able to understand and comply with protocol requirements, instructions, and any protocol-stated restrictions

   Exclusion criteria:
8. The Investigator or qualified designee considers the subject unfit for the study, based on medical interview, physical examination, or laboratory results. Individuals must be free from clinically significant illness or disease, as determined by the PI or qualified designee, with no clinically significant abnormality identified on the medical or laboratory evaluations, including 12-lead ECG
9. Positive hepatitis-B surface antigen, positive hepatitis-C, or positive HIV test
10. History of cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to screening
11. Personal or family history of medullary cell carcinoma or multiple endocrine neoplasia syndrome type 2
12. History of inadequately controlled thyroid disease, as reflected by an abnormal thyroid stimulating hormone test or free T4
13. History of gastrointestinal disease that could affect fat or bile acid ab-sorption, including inflammatory bowel disease, chronic diarrhea, Crohn's disease, or malabsorption syndromes within the past year. Note: Subjects with a cholecystectomy more than 1 year prior to screening can be considered for inclusion in the study
14. History of gastrointestinal surgical intervention for obesity
15. History of chronic or acute pancreatitis
16. History of significant drug or other allergy or hypersensitivity that, in the opinion of the Investigator or qualified designee, contraindicates the subject's participation in the study
17. History of alcohol abuse, defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is defined as equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine
18. Unwilling to abstain from alcohol from 24 hours prior to the start of dosing until discharge from the clinic
19. Smoked or used tobacco- or nicotine-containing products within the previous 6 months prior to Screening
20. Treatment with an investigational drug or participated in any other interventional clinical study during the previous 30 days or within 5 half-lives after the last dose of the investigational drug, whichever is longer. Note: 30-day/5-half-life washout is defined as last dose of investigational drug in the previous study until the first screening visit in the current study
21. Unwilling to refrain from the use of illicit drugs and unwilling to ad-here to other protocol-stated restrictions while participating in the study
22. Unwilling to abstain from caffeine- or xanthine-containing products from 24 hours prior to dosing until discharge from the clinic
23. A positive drug and alcohol screen at screening or check-in prior to dosing
24. A positive pre-study urine cotinine screen indicating use of tobacco/nicotine-containing products at Screening or check-in prior to dosing
25. Use of prescription or non-prescription drugs, vitamins, or dietary/herbal supplements within 1 week prior to the dosing of study drug through the final follow-up visit
26. Donated 500 mL or greater of blood within 56 days prior to dosing or plans on donating blood in the 30 days following completion of the study
27. Have any condition that, in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 31 days
  The primary outcome for this study is Dose Limiting Toxicity, which is the composite of any SAE, any pancreatitis(as measured by amylase) or renal dysfunction (as measured by serum creatinine)

SECONDARY OUTCOMES:
Maximum Plasma Concentration | Up to 720 hours
  Cmax
Glycosylated Hemoglobin | Up to 720 hours
  HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Lazaroff, MSN, Study Director — Gan and Lee Pharmaceuticals, USA Corp
Locations (1):
- Celerion, Lincoln, Nebraska, United States